CLINICAL TRIAL: NCT04518956
Title: Comparative Study Between the Effect of Shockwave Therapy and Low-intensity Pulsed Ultrasound (LIPUS) on Bone Healing of Mandibular Fracture
Brief Title: Shockwave Therapy Versus LIPUS on Mandibular Fracture Bone Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mandibular fracture healing
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inter maxillary fixation and exposure to shockwave therapy (Experimental)
  Interventions: Procedure: inter maxillary fixation with shockwave therapy
- Inter maxillary fixation and exposure to low intensity pulsed (Experimental)
  Interventions: Procedure: Inter maxillary fixation and exposure to low intensity pulsed
- Inter maxillary fixation only (Active Comparator)
  Interventions: Procedure: Inter maxillary fixation

INTERVENTIONS:
Procedure: inter maxillary fixation with shockwave therapy — Shockwave therapy device which give 1500-4000 pulses per session with or without anesthesia, and the treatment session takes approximately 5-10 minutes at the day after surgery.
  Arms: Inter maxillary fixation and exposure to shockwave therapy
Procedure: Inter maxillary fixation and exposure to low intensity pulsed — Low-intensity pulsed ultra sound was applied three times weekly for six weeks from the second day after surgery.
  Arms: Inter maxillary fixation and exposure to low intensity pulsed
Procedure: Inter maxillary fixation — Closed reduction will be done. Intermaxillary fixation (IMF) will be secured after proper reduction of the fractured segments to assure proper occlusion using upper and lower arch bars or eyelet wires for six weeks.
  Arms: Inter maxillary fixation only

SUMMARY:
compare between the effect of shockwave therapy and low-intensity pulsed ultrasound on healing process of fresh mandibular fractures

DETAILED DESCRIPTION:
The mandible is the commonest facial bone to fracture. Mandibular fractures represent more than 74% of all maxillofacial fractures.

To compare between the effect of shockwave therapy and low-intensity pulsed ultrasound on healing process of fresh mandibular fractures.

A total of 21 patients; aged between 20-40 years, who have mandibular fracture were selected for this study from the outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University. In this study all patients were subjected to closed reduction and intermaxillary fixation. This will be followed by shockwave therapy in seven patients as a study group and by low-intensity pulsed ultrasound in seven patients as study group. Seven patients will receive neither and will constitute the control group.

ELIGIBILITY:
Inclusion Criteria -Patients selected for this study will have fresh fracture mandible which is indicated for closed reduction.

Exclusion Criteria

-Patients having the following criteria will be excluded scars, burns, infection in the Skin in the relevant working area

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12-18 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-06-23 (Actual)

PRIMARY OUTCOMES:
Change in pain scale | after 24 hours and 1 week
  pain was scores using visual analouge scale from 0 to 10 0 means no pain 10 most severe pain
Change in bone density | after 6 Weeks and 12 weeks
  using CT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt